CLINICAL TRIAL: NCT02450630
Title: Strengthening Referral of Sick Children Form the Private Health Sector
Brief Title: Assessing the Effect of Strengthening Referral of Sick Children From the Private Health Sector and Its Impact on Referral Uptake in Uganda.
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Ministry of Health, Uganda (Other Government)
Collaborators: Makerere University (Other); Columbia University (Other); London School of Hygiene and Tropical Medicine (Other); University of Copenhagen (Other)
Responsible Party: Principal Investigator, Anthony Mbonye, Director Health Servces in charge of community and clinical services, Ministry of Health, Uganda
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: 2000004199
Record Dates: First submitted 2015-05-09; First posted 2015-05-21 (Estimated); Last update posted 2015-05-21 (Estimated); Status verified 2015-05

CONDITIONS: Malaria
MeSH Terms: conditions — Malaria

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- training on diagnosis, treatment and referral of children (Experimental): Intervention Arm : training in diagnosis, treatment and referral of sick children
  Interventions: Behavioral: Strenghtened referral of children
- Presumptive treament of sick children (No Intervention): Control Arm - Training of private providers in completing study tools i.e. filling in register and referral forms. No training in diagnosis, treatment and referral and no community awareness on referral

INTERVENTIONS:
Behavioral: Strenghtened referral of children — Community awareness on referral+ trained private providers in using RDTs/ICCM to treat and refer sick children + supervision and regular meetings between the private and public sector.All health workers in the intervention arm will be trained on how to recognize and distinguish uncomplicated & severe malaria, supplying unit-dose packaged Coartem® to customers with uncomplicated malaria, and administration of rectal artesunate pre-referral treatment and referral for sick children with severe and complicated malaria, diarrhoea and pneumonia.Private outlets in intervention arm will be trained to improve diagnosis, treatment and referral of children. The intervention will thus contribute to better health seeking practices at a community level and improved quality of care in the private sector
  Other Names: Improved referral of sick children
  Arms: training on diagnosis, treatment and referral of children

SUMMARY:
Uganda's under-five mortality is high, currently estimated at 90/1000 live births (Uganda Bureau of Statistics 2011). Poor referral of sick children that seek care from the private sector is one of the contributory factors. The proposed intervention aims to improve uptake of referral advice for children that seek care from private facilities (registered drug shops/private clinics).

The project will be implemented in Mukono district, central Uganda selected because a recent concluded trial in the district showed that drug shop vendors (DSVs) adhere to diagnostic test results, treat appropriately and refer sick children; although uptake of referral is poor. The main reasons attributed to the observed poor referral were negative attitude towards referral forms from drugs shops by the health workers at referral facilities,perceptions of poor quality of care at referral facilities and costs involved (Hutchinson. 2012; Hutchinson et al. 2013 in press)..

Thus the proposed project is a follow up to address these factors with the aim to improve uptake of referral. This project is in line with the Uganda's Health sector and USAID Mission's health priorities of strengthening the health system. Critical barriers in the implementation of child survival interventions are poor quality of care in the private sector and timely referral and uptake of referral advice at community level. These barriers may be attributed to inadequate training of providers in the private sector (in diagnosis and management of childhood illnesses); inadequate supervision and regulation; poor linkages and collaboration between the public and private sectors; and non-existent linkages between community structures and the private sector. The barriers will be addressed through an intervention with three components; i) VHTs will be trained to do community sensitization and initiate community discussions aimed at identifying community support mechanisms for financial hardship (to be community led and managed) - e.g. communities to be encouraged to establish community credit/insurance schemes for referral VHTs will register children and facilitate follow up of sick children ii) supervision of providers in the private sector to diagnose, treat and refer sick children, iii) regular meetings between the public and private providers (convened by the district health team) to discuss the referral system.

DETAILED DESCRIPTION:
Research Questions/Goals and Specific Objectives:

Research question: The study aims to answer the question whether integrated intervention of VHT registration of children (registration of children will enable follow up by VHTs), community sensitization and regular meetings between the public and private providers on referral of sick children targeting women and men is cost-effective and can improve uptake of referral advice.

Goal: The goal of the study is to assess the effect of a strengthened referral system from the private sector on uptake of referral advice and its cost-effectiveness. The project addresses poor referral of children as one of the challenges in the reduction of under-five mortality in Uganda.

Primary objective:

1. To asses the effect of strengthening the referral system on uptake of referral of sick children who seek care in the private sector.

Secondary objectives

1. To explore factors which influence the referral or non-referral of sick children from the private sector.
2. To assess the cost effectiveness of uptake of referral of sick children who seek care in the private sector.

   Uganda's under-five mortality is high, currently estimated at 90/1000 live births (UDHS, 2011) Poor referral of sick children that seek care from the private sector is one of the contributory factors. Previous studies in Uganda and elsewhere have found out that referral of sick children to higher levels of care is poor (Oryema, 2009, Achan et al 2011; Font et al 2002, Kallander et al 2006 ), In Uganda several studies have estimated referral of children to be as low as 8% (Kallander et al 2006) to 28% (Peterson et al 2004). Several factors have been attributed to the poor referral like long distances to health facilities, high costs involved in referral, poor attitudes of health workers, lack of drugs at health facilities and lack of involvement of fathers in the referral process (Mbonye 2003, Font et al 2002).

   A study in Uganda found that of the 70% of patients who sought treatment at private clinics within 1 week of onset of symptoms only 7% were properly managed (treated according to National Guidelines). The study concluded that at private facilities possible strategies include training and social marketing of prepackaged treatment for STDs (Jacobs et al 2004).

   In Tanzania, it has been found that in urban private-sector clinics, flexible clinics hours, prompt services, and efforts to improve respect, privacy and confidentiality may prove more helpful in increasing visit adherence (Miller et al 2014).

   The proposed intervention aims to improve referral and uptake of referral advice of children that seek care from private facilities by addressing constraints to the referral of children. The private sector providers participating in this project will include private clinics and registered drug shops. A recently concluded trial has shown that staff in drug shops were mainly female, of whom over 50% were qualified health workers (state enrolled nurse or above). The majority of drug shop vendors had received no prior training on malaria case management, and had little knowledge at baseline of ACT as the first-line anti-malarial drug, or what an mRDT was used for (Mbonye et al. submitted, 2014).

   The project will be implemented in Mukono District, Central Uganda. There is a high prevalence of diarrhea (22.3%), acute respiratory tract infection (12%) and fever (42%) among children aged <5 years (Uganda Bureau of Statistics 2011).

   This district has been selected because of a recent concluded trial showed drug shop vendors (DSVs) adhere to malaria diagnostic test results, treat appropriately and refer sick children; although uptake of referral is poor. Thus proposed project therefore is a follow up to assess factors that lead to poor uptake of referral.

   The main focus of this project is to implement a community-based intervention to encourage uptake of referral. This is because non-compliance or delayed uptake of referral threatens child survival. The project targets children aged less than five years, especially in rural areas who have poor access to health interventions. Three of the barriers to effective treatment are poor quality of care in the private sector, timely referral, and uptake of referral advice at a community level . Poor quality of care in the private sector may be attributed to inadequate training of providers in the private sector (in diagnosis and management of childhood illnesses); inadequate supervision and regulation; poor linkages and collaboration between the public and private sectors. Poor uptake of referral advice may be due to lack of awareness of severe signs for childhood illnesses and their consequences; and poor preparation of household's especially inadequate male involvement in child care; and non-existent linkages between community structures and the public-private sectors. The cost-effectiveness and sustainability of such innovative ways to scale up interventions is not known.

   The proposed research will be implemented in a district endemic for malaria, pneumonia and diarrhea with both peri-urban and rural areas. It has numerous registered drug shops and private clinics that are capable of diagnosing febrile illnesses with RDTs and treat malaria appropriately and refer sick children (Mbonye et al 2013, submitted). The target population is children with febrile illness who seek treatment at private outlets. It is hypothesized that raising community awareness targeting households (women and spouses) and initiating discussion on saving schemes for referral costs will lead to completion of referral advice for sick children. The intervention will be supported with qualitative studies to explore reasons for uptake of referral or not; and lessons for policy action. The contextual issues to be explored by the qualitative research will include involvement of community structures (VHTs) in raising awareness, the modalities of linkages between the community and public-private health facilities, and incentives for referral.

   The first aspect of innovation is using VHTs to register children and do community sensitization. The second innovation in this project is introducing integrated management of malaria, pneumonia and diarrhea in private outlets, that has been only implemented at community level and in health facilities. The third aspect of innovation is to involve the private sector in the referral of sick children. Understanding the referral system is a new research area that could inform the private-public interactions with wider public health implications for child survival.

   There will be meetings convened by the district health system between private and public providers in the study communities to introduce the study and discuss the referral process. Referral forms will be developed and discussed with all stakeholders; as well as SOPs for handling referral cases. In the previous trial of RDTs in drug shops in Mukono district, referral forms were in the local language and health workers despised them. In this present study the investigators shall modify them and pilot forms in English, and put in place supporting interventions to foster acceptance of referrals from the private sector.

   The third aspect of innovation is to involve VHTs, an established community structure ( MOH, 1999; MOH 2010) to register all children aged less than 5 years, distribute health education materials and enlist male heads of households and women to be active in the care and referral of children. Since men are crucial in decision making and control of resources, the investigators hypothesize that this innovation is likely to improve timely referral and uptake of referral advice. VHTs currently have no collaboration with the private sector thus creating links between VHTs and the private sector is creative and is likely to provide lessons for future scale up of health interventions. Meetings between the private and public providers have never taken place and establishing such interaction would be innovative.

   The immediate sustainable impact will be appropriate treatment of sick children. The long term effect is reduction in child mortality, which may lead to reduction in fertility as women would embrace more family planning methods once the survival of children improves. The potential scientific impact of the project will be evaluated by capturing data on referrals, where sick children are referred, uptake of the referral compared between the two arms.
3. Objectives & Outcome Measure(s) A. Study objectives

Primary objective:

1. To assess the effect of strengthening the referral system on uptake of referral of sick children who seek care in the private sector.

Secondary objectives

1. To explore factors which influence the referral or non-referral of sick children from the private sector.
2. To assess the cost-effectiveness of timely and uptake of referral of sick children seen in the private sector.

B. Study Outcome measure(s) List and describe the primary outcome measure and if applicable, secondary outcome measures including both quantitative and qualitative outcomes. Discuss the validity of the selected outcome(s). Provide evidence that selected outcomes will provide relevant, valid, and reliable measures of all study objectives.

The primary outcome:

• The proportion of sick children referred from the private sector that completes the referral process (seen at higher health facilities).

Co-primary outcomes:

* Appropriate case management for malaria, pneumonia and diarrhea among children in the private sector.
* The cost-effectiveness of timely and uptake of referral of sick children.

Secondary outcomes:

* The proportion of sick children seeking care at private outlets within 24 hours of onset of symptoms
* The time between consultations at private outlets and uptake of referral at health facilities (referral facilities)
* The proportion of sick children receiving prompt appropriate treatment from a private sector outlet.
* Factors which influence the referral or non-referral of sick children from the private sector.

All private outlets in both arms will be trained to record data on sick children aged less than 5years who seek care at private outlets:

1. Demographic (age, sex, relationship to caretaker, marital status of caretaker, education levels, rural/urban residence)
2. Social-economic data (household income, ownership of household items that determine expenditure and consumption levels, address and telephone contacts of caretakers));
3. Type of illnesses, treatment given, prescription of drugs, referral advice, children referred and where referred.

These data will be captured in patient registers and treatment forms distributed in the intervention and control clusters.

ELIGIBILITY:
Inclusion Criteria:

* A cluster is defined to be a parish or neighboring parishes if the distance between any two private outlets located in each of the parishes is<1 km( to minimize possible spill over).
* Any of the 63 parishes/clusters in Mukono district will be eligible if:

  i) Contain more than 200 households to ensure a sufficient number of sick children visiting the private outlets

ii) Contained at least one registered drug shop/private clinic with the district drug inspector (DDI).

iii) Contain a health centre II, the lowest public health facility where early treatment is sought.

Exclusion Criteria:

i) Unregistered drug shop/private clinic

ii) No HFII government health facility located within the same parish

iii) Fewer than 200 households in the parish where drug shop/private clinic is located

iv) If the health facility does not have a qualified health worker. Some government health HCIIs in Uganda are run by nursing aides.

Max Age: 5 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 8910 (Estimated)
Dates: Start 2015-05; Primary Completion 2016-12 (Estimated); Study Completion 2017-05 (Estimated)

PRIMARY OUTCOMES:
The proportion of sick children referred from the private sector that complete the referral process (seen at higher level facilities). | 2 years
  This will be measured as a proportion of referred sick children of the total number of sick children

SECONDARY OUTCOMES:
The proportion of sick children seeking care and receiving prompt treatment at private outlets within 24 hours of onset of symptoms; | 2 years
  Measured as the number of children seen at private facilities within 24 hours of the total number of sick children
The time between consultations at private outlets and uptake of referral at health facilities (referral facilities); | 2 years
  measure by time in hours
The cost-effectiveness of the intervention | 2years
  The costs and effectiveness of the intervention per arm will be calculated as incremental cost per Disability Adjusted Life Years (DALY) averted of introducing a strengthened referral system (the cost-effectiveness)

CONTACTS AND LOCATIONS:
Overall Officials: Anthony K Mbonye, PhD, Principal Investigator — Minstry of Health Uganda

REFERENCES:
- [Derived] Mbonye AK, Buregyeya E, Rutebemberwa E, Lal S, Clarke SE, Hansen KS, Magnussen P, LaRussa P. Treatment of Sick Children Seeking Care in the Private Health Sector in Uganda: A Cluster Randomized Trial. Am J Trop Med Hyg. 2020 Mar;102(3):658-666. doi: 10.4269/ajtmh.19-0367. PMID 31971139
- [Derived] Buregyeya E, Rutebemberwa E, LaRussa P, Mbonye A. Strengthening referral of sick children from the private health sector and its impact on referral uptake in Uganda: a cluster randomized controlled trial protocol. BMC Health Serv Res. 2016 Nov 11;16(1):646. doi: 10.1186/s12913-016-1885-5. PMID 27835980